CLINICAL TRIAL: NCT02716870
Title: Effect of Important Food Sources of Fructose-containing Sugars on Cardiometabolic Risk Factors: A Series of Systematic Reviews and Meta-analyses of Controlled Trials to Inform Dietary Guidelines, Public Health Policy, and Future Trial Design
Brief Title: Meta-analyses of the Effect of Important Food Sources of Sugars on Cardiometabolic Risk Factors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Canadian Diabetes Association (Other); The Physicians' Services Incorporated Foundation (Other); Banting & Best Diabetes Centre (Other)
Responsible Party: Principal Investigator, John Sievenpiper, Associate Professor, University of Toronto
Other Study IDs: CDA-Sugars 2015
Record Dates: First submitted 2016-03-02; First posted 2016-03-23 (Estimated); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Dyslipidemia; Diabetes; Prediabetes; Dysglycemia; Gout; Hypertension; Non-alcoholic Fatty Liver Disease; Cardiovascular Disease
Keywords: Systematic review and meta-analysis; Evidence-based medicine (EBM); Evidence-based nutrition (EBN); Clinical practice guidelines; Clinical trials; Dietary sugars; Fructose; High fructose corn syrup; Fruit; Isocaloric; Hypercaloric; Cardiometabolic risk factors; Triglycerides; Cholesterol; Glycemic control; Insulin resistance; Body weight; Uric acid; Blood pressure; Fatty liver; Fasting; Postprandial
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus; Prediabetic State; Gout; Hypertension; Non-alcoholic Fatty Liver Disease; Cardiovascular Diseases; Insulin Resistance; Body Weight; Fatty Liver; Fasting | interventions — Fructose; Sucrose; High Fructose Corn Syrup; Honey

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Fructose-containing Sugars — An intervention in which calories from fructose-containing sugars are substituted, added, or subtracted in the diet
  Other Names: fructose, sucrose, high-fructose corn syrup (HFCS), honey

SUMMARY:
Fructose-containing sugars have been implicated in the epidemics of obesity, diabetes and related cardiometabolic disorders. This view is supported by lower quality evidence from ecological observations, animal models, and select human trials. Higher level evidence from controlled trials and prospective cohort studies have been inconclusive. Whether sugars contribute to cardiometabolic complications independent of their calories remains unclear. To address the uncertainties, the investigators propose to conduct a series of systematic reviews and meta-analyses of the totality of the evidence from controlled trials to distinguish the contribution of fructose-containing sugars from that of energy in the development of markers of cardiometabolic risk. The findings generated by this proposed knowledge synthesis will help improve the health of consumers through informing evidence-based guidelines and improving health outcomes by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

DETAILED DESCRIPTION:
Background: Sugars have emerged as one of the most important public health concerns. Attention has focused particularly on fructose-containing sugars (fructose, sucrose, high fructose corn syrup, honey, etc), which collectively have been indicted as drivers of various cardiometabolic complications. This special view rests on the unique metabolic and endocrine responses to fructose. Unlike glucose, fructose is thought to bypasses negative feedback controls acting as an unregulated substrate for de novo lipogenesis and impair satiety signaling resulting in weight gain. In support of these mechanisms, animal models, low-quality ecological studies, and select human trials of overfeeding at levels of exposure far beyond population intakes have reported adverse metabolic effects of sugars. Higher level evidence from systematic reviews and meta-analyses of controlled trials, however, suggests that any effects of sugars are mediated by excess calories rather than the sugars per se. It remains unclear whether fructose-containing sugars contribute to cardiometabolic complications independent of their calories.

Need for proposed research: High quality systematic reviews and meta-analyses of controlled trials represent the highest level of evidence to support dietary guidelines and public health policy development. As dietary guidelines and public health policy have shifted toward food and dietary-pattern based recommendations, there is an urgent need for systematic reviews and meta-analyses comparing the role of different food sources of sugars in the development of cardiometabolic diseases.

Objective: The investigators will conduct a series systematic reviews and meta-analyses to distinguish the effect of fructose-containing sugars from that of energy on measures of cardiometabolic risk in controlled trials.

Design: Each systematic review and meta-analysis will be conducted according to the Cochrane Handbook for Systematic Reviews of Interventions and reported according to the Preferred Reporting Items for Systematic Reviews and Meta-Analyses (PRISMA).

Data sources: MEDLINE, EMBASE, and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms supplemented by hand searches of references of included studies.

Study selection: The investigators will include randomized and non-randomized controlled trials >= 7-days in duration to assess the effect of fructose-containing sugars (fructose, sucrose, high fructose corn syrup, honey, etc) on measures of cardiometabolic risk. To allow for the separation of the effect of sugars from that of energy, 4 trial designs will be considered: (1) 'substitution' trials, in which fructose-containing sugars added to foods and beverages are compared with other macronutrient sources (usually starch or other sugars) under energy matched conditions; (2) 'addition' trials, in which fructose-containing sugars supplement a diet with excess energy compared to the same diet alone without the excess energy; (3) 'subtraction' trials, in which energy from fructose-containing sugars (usually in the form of sugars-sweetened beverages) is reduced by displacing it with water and/or no-calorie or low-calorie sweeteners or by eliminating it altogether from the background diet; and (4) 'ad libitum' trials, in which energy from fructose-containing sugars are freely replaced with other sources of energy (usually complex carbohydrates or fat) without any strict control of either the study foods or the background diet. Trials will be categorized by sources of fructose-containing sugars (fruits, fruit juices, sugars-sweetened beverages, liquid meal replacements, dairy products, sweets/desserts/baked goods, mixed sources) and chi squared tests will be used to determine between-group differences.

Data extraction: Two or more investigators will independently extract relevant data and assess risk of bias using the Cochrane Risk of Bias Tool. All disagreements will be resolved by consensus. Standard computations and imputations will be used to derive missing variance data.

Outcomes: Five sets of outcomes will be assessed: (1) glycemic control (glycated blood proteins [HbA1c, fructosamine, glycated albumin], fasting glucose, and fasting insulin), (2) blood lipids (Established therapeutic lipid targets [LDL-cholesterol, non-HDL-cholesterol, apolipoprotein B (apo B), HDL-cholesterol, triglycerides]), (3) blood pressure (systolic blood pressure and diastolic blood pressure), (4) uric acid, (5) non-alcoholic fatty liver disease (NAFLD) (intrahepatocellular lipids [IHCL], alanine aminotransferase [ALT], aspartate aminotransferase [AST]) and inflammation (c-reactive protein [CRP], IL-6, TNF-alpha).

Data synthesis: Mean differences will be pooled using the generic inverse variance method for each food source of fructose-containing sugars. Random-effects models will be used even in the absence of statistically significant between-study heterogeneity, as they yield more conservative summary effect estimates in the presence of residual heterogeneity. Fixed-effects models will only be used where there is <5 included studies. Paired analyses will be applied for crossover trials. Heterogeneity will be assessed by the Cochran Q statistic and quantified by the I2 statistic. To explore sources of heterogeneity, the investigators will conduct sensitivity analyses, in which each study is systematically removed. If there are >=10 studies, then the investigators will also explore sources of heterogeneity by a priori subgroup analyses by age (children [=<18 years of age], adults), health status (metabolic syndrome criteria, diabetes, overweight/ obese, healthy), comparator type, fructose- containing sugar form (sucrose, high fructose corn syrup [HFCS], honey, fructose), dose (=<10% energy, >10%), baseline measurements, randomization, study design (parallel, crossover), energy balance (positive, neutral, negative), follow-up (<8-weeks, >=8-weeks), feeding control (metabolic, supplemented, dietary advice), funding (agency, industry, agency+industry, not reported), and risk of bias. Meta-regression analyses will assess the significance of categorical and continuous subgroups analyses. When >=10 studies are available, publication bias will be investigated by inspection of funnel plots and formal testing using the Egger and Begg tests. If publication bias is suspected, then the investigators will attempt to adjust for funnel plot asymmetry by imputing the missing study data using the Duval and Tweedie trim and fill method.

Evidence Assessment: The strength of the evidence for each outcome will be assessed using the Grading of Recommendations Assessment, Development and Evaluation (GRADE).

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition, diabetes, obesity, and cardiovascular disease. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined. Applicant/Co-applicant Decision Makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

Significance: The proposed project will aid in knowledge translation related to the role of dietary fructose-containing sugars and important food sources of these sugars in the development of cardiometabolic diseases, strengthening the evidence-base for guidelines and improving health outcomes by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

ELIGIBILITY:
Inclusion Criteria:

* Trials in humans
* Oral fructose-containing sugars intervention
* Presence of an adequate comparator (substitution, addition, subtraction, or ad libitum control)
* Diet duration >=7 days
* Viable outcome data

Exclusion Criteria:

* Non-human trials
* Observational studies
* IV or parenteral fructose-containing sugars
* Lack of suitable comparator (i.e. a comparator arm that contains substantial fructose-containing sugars)
* Diet duration <7 days
* No viable outcome data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals, both children and adults, regardless of health status.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control | Up to 20 years
  glycated blood proteins, fasting blood glucose, fasting blood insulin
Established Therapeutic Blood Lipid Targets | Up to 20 years
  LDL-cholesterol, apol B, non-HDL-cholesterol, HDL-cholesterol, triglycerides
Blood Pressure | Up to 20 years
Uric Acid | Up to 20 years
  Blood uric acid concentrtaions
Non-Alcoholic Fatty Liver Disease (NAFLD) | Up to 20 years
  Intrahepatocellular lipid concentrations (IHCL), ALT
Inflammation | Up to 20 years
  c-reactive protein (CRP)

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD,PhD,FRCPC, Principal Investigator — University of Toronto
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Sievenpiper JL, de Souza RJ, Mirrahimi A, Yu ME, Carleton AJ, Beyene J, Chiavaroli L, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Kendall CW, Jenkins DJ. Effect of fructose on body weight in controlled feeding trials: a systematic review and meta-analysis. Ann Intern Med. 2012 Feb 21;156(4):291-304. doi: 10.7326/0003-4819-156-4-201202210-00007. PMID 22351714
- [Background] Ha V, Sievenpiper JL, de Souza RJ, Chiavaroli L, Wang DD, Cozma AI, Mirrahimi A, Yu ME, Carleton AJ, Dibuono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ. Effect of fructose on blood pressure: a systematic review and meta-analysis of controlled feeding trials. Hypertension. 2012 Apr;59(4):787-95. doi: 10.1161/HYPERTENSIONAHA.111.182311. Epub 2012 Feb 13. PMID 22331380
- [Background] Cozma AI, Sievenpiper JL, de Souza RJ, Chiavaroli L, Ha V, Wang DD, Mirrahimi A, Yu ME, Carleton AJ, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ. Effect of fructose on glycemic control in diabetes: a systematic review and meta-analysis of controlled feeding trials. Diabetes Care. 2012 Jul;35(7):1611-20. doi: 10.2337/dc12-0073. PMID 22723585
- [Background] Chiavaroli L, de Souza RJ, Ha V, Cozma AI, Mirrahimi A, Wang DD, Yu M, Carleton AJ, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ, Sievenpiper JL. Effect of Fructose on Established Lipid Targets: A Systematic Review and Meta-Analysis of Controlled Feeding Trials. J Am Heart Assoc. 2015 Sep 10;4(9):e001700. doi: 10.1161/JAHA.114.001700. PMID 26358358
- [Background] Wang DD, Sievenpiper JL, de Souza RJ, Chiavaroli L, Ha V, Cozma AI, Mirrahimi A, Yu ME, Carleton AJ, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ. The effects of fructose intake on serum uric acid vary among controlled dietary trials. J Nutr. 2012 May;142(5):916-23. doi: 10.3945/jn.111.151951. Epub 2012 Mar 28. PMID 22457397
- [Background] Chiu S, Sievenpiper JL, de Souza RJ, Cozma AI, Mirrahimi A, Carleton AJ, Ha V, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Don-Wauchope AC, Beyene J, Kendall CW, Jenkins DJ. Effect of fructose on markers of non-alcoholic fatty liver disease (NAFLD): a systematic review and meta-analysis of controlled feeding trials. Eur J Clin Nutr. 2014 Apr;68(4):416-23. doi: 10.1038/ejcn.2014.8. Epub 2014 Feb 26. PMID 24569542
- [Derived] Liu Q, Chiavaroli L, Ayoub-Charette S, Ahmed A, Khan TA, Au-Yeung F, Lee D, Cheung A, Zurbau A, Choo VL, Mejia SB, de Souza RJ, Wolever TMS, Leiter LA, Kendall CWC, Jenkins DJA, Sievenpiper JL. Fructose-containing food sources and blood pressure: A systematic review and meta-analysis of controlled feeding trials. PLoS One. 2023 Aug 15;18(8):e0264802. doi: 10.1371/journal.pone.0264802. eCollection 2023. PMID 37582096
- [Derived] Qi X, Chiavaroli L, Lee D, Ayoub-Charette S, Khan TA, Au-Yeung F, Ahmed A, Cheung A, Liu Q, Blanco Mejia S, Choo VL, de Souza RJ, Wolever TMS, Leiter LA, Kendall CWC, Jenkins DJA, Sievenpiper JL. Effect of Important Food Sources of Fructose-Containing Sugars on Inflammatory Biomarkers: A Systematic Review and Meta-Analysis of Controlled Feeding Trials. Nutrients. 2022 Sep 26;14(19):3986. doi: 10.3390/nu14193986. PMID 36235639
- [Derived] Ayoub-Charette S, Chiavaroli L, Liu Q, Khan TA, Zurbau A, Au-Yeung F, Cheung A, Ahmed A, Lee D, Choo VL, Blanco Mejia S, de Souza RJ, Wolever TM, Leiter LA, Kendall CW, Jenkins DJ, Sievenpiper JL. Different Food Sources of Fructose-Containing Sugars and Fasting Blood Uric Acid Levels: A Systematic Review and Meta-Analysis of Controlled Feeding Trials. J Nutr. 2021 Aug 7;151(8):2409-2421. doi: 10.1093/jn/nxab144. PMID 34087940
- [Derived] Choo VL, Viguiliouk E, Blanco Mejia S, Cozma AI, Khan TA, Ha V, Wolever TMS, Leiter LA, Vuksan V, Kendall CWC, de Souza RJ, Jenkins DJA, Sievenpiper JL. Food sources of fructose-containing sugars and glycaemic control: systematic review and meta-analysis of controlled intervention studies. BMJ. 2018 Nov 21;363:k4644. doi: 10.1136/bmj.k4644. PMID 30463844